CLINICAL TRIAL: NCT06257823
Title: Exploring Vascular Contributions to Cognitive Decline and Dementia
Brief Title: Vascular Cognitive Decline and Dementia
Acronym: ENIGMA
Status: Recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Janne Kaergard Mortensen, Associate Professor, MD, PhD, Aarhus University Hospital
Other Study IDs: 1-10-72-253-20
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
Keywords: Dementia; Cognitive impairment; MRI; Extracellular vesicles; Stroke
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Dementia; Cognitive Dysfunction; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The ENIGMA study is a single-centre prospective clinical observational study with the aim to investigate vascular contributions to cognitive decline and dementia. By studying MRI-defined capillary dysfunction and EV profiles, the ENIGMA study links novel imaging and basic research techniques to a clinical cohort of stroke patients. With this study we hope to enhance the understanding of the mechanisms behind post-stroke cognitive decline and dementia.

DETAILED DESCRIPTION:
Post-stroke cognitive impairment (PSCI) is common. However, the underlying pathophysiology remains largely unknown. Understanding how microvascular changes relate to PSCI and finding markers that can predict PSCI, could be a first step towards better screening and management.

Cerebral capillary dysfunction is characterized by limited oxygen extraction from the brain capillaries due to age- and risk factor-related capillary flow heterogeneity. Capillary dysfunction is a pathophysiological feature of cerebral small vessel disease (cSVD) and may play an important role in the vascular mechanisms underlying PSCI. Extracellular vesicles (EVs) carry molecules between cells. EV profiles may change during acute stroke, in the chronic stroke phase, and according to the level of cSVD, and EV profiles may therefore act as disease biomarkers.

The ENIGMA study aims to investigate capillary dysfunction and EV profiles as predictors of cognitive function one year after acute ischemic stroke (AIS) and transient ischemic attack (TIA). Consecutive patients with AIS and TIA are included and followed for one year with follow-up visits at three and 12 months. An MRI is performed at 24 hours and 12 months after admission. EV profiles will be characterised from blood samples drawn at 24 hours and three months after admission. Cognitive function is assessed three and 12 months after AIS and TIA using the Repeatable Battery for the Assessment of Neuropsychological Status and the Montreal Cognitive Assessment (MoCA).

The study has two main objectives: 1) to study associations between capillary dysfunction and PSCI and 2) to assess associations between EV profiles and PSCI.

ELIGIBILITY:
Inclusion Criteria:

* AIS or TIA with a clinically relevant diffusion restriction identified on MRI DWI-sequence on admission
* Admittance within 24 hours from symptom onset
* Age ≥ 60

Exclusion Criteria:

* Dependency in activities of daily living (mRS score > 2)
* Known dementia, neurodegenerative disease, or other significant brain disease
* Concomitant life-threatening disease
* Contraindications to undergo MRI
* Allergy or intolerance to MRI contrast agents
* eGFR < 30
* Unable to give written informed consent
* Deemed unfit for follow-up

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 60 years admitted with AIS or TIA to the comprehensive stroke center at Aarhus University Hospital within 24 hours of symptom onset.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Post-stroke cognitive decline | 12 months
  Change in RBANS index score from three to 12 months follow-up
Post-stroke cognitive impairment | 12 months
  Total RBANS index score

SECONDARY OUTCOMES:
Post-stroke cognitive decline | 12 months
  Change in MoCA score from three to 12 months follow-up
Post-stroke cognitive impairment | 12 months
  MoCA score at 12 months follow-up
Post-stroke depression | 12 months
  Measured on the major depression inventory
Physical activity | 12 months
  Measured on the Physical Activity Scale for the Elderley

CONTACTS AND LOCATIONS:
Overall Officials: Janne Kaergaard Mortensen, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All investigators will have access to the entire dataset. Trial metadata, including, but not limited to codebooks, data dictionaries and analysis code will be shared on a repository under a permissive license. Upon completing a collaboration agreement, individual patient trial data may be shared upon reasonable request. Patient data will not be made publicly available.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Not decided
Access Criteria: Upon completing a collaboration agreement, individual patient trial data may be shared upon reasonable request. Patient data will not be made publicly available.

REFERENCES:
- [Derived] Vestergaard SB, Damsbo AG, Pedersen NL, Zachariassen K, Drasbek KR, Ostergaard L, Andersen G, Dalby RB, Mortensen JK. Exploring vascular contributions to cognitive impairment and dementia (ENIGMA): protocol for a prospective observational study. BMC Neurol. 2024 Apr 3;24(1):110. doi: 10.1186/s12883-024-03601-7. PMID 38570800